CLINICAL TRIAL: NCT00246025
Title: A Randomised, Parallel-group, Double-blind, Placebo Controlled Study to Investigate the Efficacy and Safety of BIBR 1048 in Prevention of Venous Thromboembolism in Patients With Primary Elective Total Knee Replacement Surgery
Brief Title: A Study of BIBR 1048 in Prevention of Venous Thromboembolism in Patients With TKR Surgery.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1160.50
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2010-12-17 (Estimated); Last update posted 2014-06-09 (Estimated); Status verified 2014-02

CONDITIONS: Arthroplasty, Replacement, Knee; Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Dabigatran

ARMS (4):
- Dabigatran etexilate 110 mg (Experimental): Dabigatran etexilate 110 mg capsule, once a day, oral administration
  Interventions: Drug: Dabigatran etexilate
- Dabigatran etexilate 150 mg (Experimental): Dabigatran etexilate 150 mg capsule, once a day, oral administration
  Interventions: Drug: Dabigatran etexilate
- Dabigatran etexilate 220 mg (Experimental): Dabigatran etexilate 110 mg capsule, 2capsules, once a day, oral administration
  Interventions: Drug: Dabigatran Etexilate
- Placebo (Placebo Comparator): matching placebo capsule, once a day, oral administration
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: Dabigatran etexilate — Dabigatran etexilate 110 mg capsule, once a day, oral administration
  Arms: Dabigatran etexilate 110 mg
Drug: Dabigatran etexilate — Dabigatran etexilate 150 mg capsule, once a day, oral administration
  Arms: Dabigatran etexilate 150 mg
Drug: Dabigatran Etexilate — Dabigatran etexilate 220 mg capsule, once a day, oral administration
  Arms: Dabigatran etexilate 220 mg
Drug: placebo — matching placebo capsule, once a day, oral administration
  Arms: Placebo

SUMMARY:
The goal of this study is to evaluate the comparative efficacy and safety of three different doses ( 110 mg, 150 mg, 220 mg) of BIBR 1048 (Dabigatran etexilate) orally, compared to placebo, in prevention of venous thromboembolism in patient with primary elective total knee replacement surgery, and to evaluate dose-response.

ELIGIBILITY:
Inclusion criteria Inclusion criteria

1. Patients scheduled to undergo a primary, unilateral elective total knee replacement
2. Male or Female 20 years of age or order
3. Patients weighing at least 40 kg
4. Written informed consent prior to the start of study participation

Exclusion criteria Exclusion criteria

1. History of bleeding diathesis
2. Constitutional or acquired coagulation disorders that in the investigator's judgment puts the patient at excessive risk for bleeding
3. Major surgery or trauma (e.g. hip fracture) within the last 3 months
4. Recent unstable cardiovascular disease, such as uncontrolled hypertension at the time of enrollment (investigator's judgment) or history of myocardial infarction within the last 3 months
5. Any history of hemorrhagic stroke or any of the following intracranial pathologies: bleeding, neoplasm, AV (arteriovenous) malformation or aneurysm or recent bleeding history
6. Condition requiring anti-coagulant therapy
7. Elevated AST(Aspartate Aminotransferase) , ALT(Alanine Aminotransferase), or any history of clinically relevant liver disease
8. Patients with a history of clinically significant renal diseases or with elevated creatinine values

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 512 (Actual)
Dates: Start 2005-10; Primary Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (38):
- Japan (38):
  - 1160.50.001 Boehringer Ingelheim Investigational Site, Eniwa, Hokkaido
  - 1160.50.018 Boehringer Ingelheim Investigational Site, Fukuoka, Fukuoka
  - 1160.50.008 Boehringer Ingelheim Investigational Site, Hachioji, Tokyo
  - 1160.50.006 Boehringer Ingelheim Investigational Site, Hirosaki, Aomori
  - 1160.50.026 Boehringer Ingelheim Investigational Site, Hiroshima, Hiroshima
  - 1160.50.011 Boehringer Ingelheim Investigational Site, Iida, Nagano
  - 1160.50.024 Boehringer Ingelheim Investigational Site, Izumisano, Osaka
  - 1160.50.045 Boehringer Ingelheim Investigational Site, Izunokuni,Shizuoka
  - 1160.50.022 Boehringer Ingelheim Investigational Site, Kagoshima, Kagoshima
  - 1160.50.027 Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - 1160.50.032 Boehringer Ingelheim Investigational Site, Kawasaki, Kanagawa
  - 1160.50.041 Boehringer Ingelheim Investigational Site, Kitakyusyu, Fukuoka
  - 1160.50.039 Boehringer Ingelheim Investigational Site, Koshigaya,Saitama
  - 1160.50.037 Boehringer Ingelheim Investigational Site, Kurume ,Fukuoka
  - 1160.50.038 Boehringer Ingelheim Investigational Site, Kurume ,Fukuoka
  - 1160.50.013 Boehringer Ingelheim Investigational Site, Kyoto, Kyoto
  - 1160.50.036 Boehringer Ingelheim Investigational Site, Matsue, Shimane
  - 1160.50.042 Boehringer Ingelheim Investigational Site, Miyazaki, Miyazaki
  - 1160.50.028 Boehringer Ingelheim Investigational Site, Musashimurayama, Tokyo
  - 1160.50.005 Boehringer Ingelheim Investigational Site, Obihiro, Hokkaido
  - 1160.50.030 Boehringer Ingelheim Investigational Site, Okayama, Okayama
  - 1160.50.021 Boehringer Ingelheim Investigational Site, Omura, Nagasaki
  - 1160.50.014 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.50.015 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.50.016 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.50.033 Boehringer Ingelheim Investigational Site, Osaka, Osaka
  - 1160.50.031 Boehringer Ingelheim Investigational Site, Saga, Saga
  - 1160.50.009 Boehringer Ingelheim Investigational Site, Sagamihara, Kanagawa
  - 1160.50.002 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1160.50.004 Boehringer Ingelheim Investigational Site, Sapporo, Hokkaido
  - 1160.50.020 Boehringer Ingelheim Investigational Site, Sasebo, Nagasaki
  - 1160.50.025 Boehringer Ingelheim Investigational Site, Sasebo, Nagasaki
  - 1160.50.034 Boehringer Ingelheim Investigational Site, Sendai, Miyagi
  - 1160.50.029 Boehringer Ingelheim Investigational Site, Shinjuku-ku,Tokyo
  - 1160.50.043 Boehringer Ingelheim Investigational Site, Shizuoka, Shizuoka
  - 1160.50.044 Boehringer Ingelheim Investigational Site, Sumida-ku, Tokyo
  - 1160.50.023 Boehringer Ingelheim Investigational Site, Tomigusuku, Okinawa
  - 1160.50.040 Boehringer Ingelheim Investigational Site, Tsukuba , Ibaraki

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Group With Placebo: Patients were treated with matching Placebo.
- Dabigatran Etexilate 110 mg: Patients were treated with 110mg dabigatran etexilate once daily.
- Dabigatran Etexilate 150 mg: Patients were treated with 150mg dabigatran etexilate once daily.
- Dabigatran Etexilate 220 mg: Patients were treated with 220mg dabigatran etexilate once daily.
Period: Overall Study
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Started | 124 | 133 | 126 | 129
Completed | 114 | 124 | 116 | 116
Not Completed | 10 | 9 | 10 | 13
Not completed — Adverse Event | 7 | 9 | 9 | 10
Not completed — Withdrawal by Subject | 3 | 0 | 1 | 2
Not completed — unsuitable medical history was found | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg | Total
Number analyzed (Participants) | 124 | 133 | 126 | 129 | 512
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.5) | 71.3 (7.9) | 70.9 (7.7) | 72.7 (6.8) | 71.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 106 | 105 | 109 | 425
  Male | 19 | 27 | 21 | 20 | 87

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Have a Composite Endpoint Consisting of Total Venous Thromboembolic Event (VTE) and All Cause Mortality During the Treatment Period.
Description: number of participants with the composite endpoint (total Venous Thromboembolic Event (VTE) and all cause mortality
Time Frame: 2 weeks study medication
Population: Full analysis set (FAS) - Full analysis set includes all patients who were randomly assigned to the treatment, received at least one oral dose, went through surgery, had an evaluable venogram for distal and proximal DVT, or had confirmed symptomatic DVT or PE, or died.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 101 | 106 | 104 | 96
percentage of participants | 56.4 | 39.6 | 32.7 | 24
Statistical Analysis 1: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; Superiority of dabigatran etexilate to placebo was tested by means of hierarchical tests. Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Test type: Superiority or Other; p = 0.0155, normal approximation method — Multiplicity was not adjusted because of hierarchical testing from highest to lowest dose; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -16.8, 95% CI [-30.2 to -3.4] — The risk differences are calculated as risk in the dabigatran groups minus risk in the placebo group
Statistical Analysis 2: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0006, normal approximation method — Multiplicity was not adjusted because of hierarchical testing from highest to lowest dose; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -23.7, 95% CI [-37.0 to -10.5] — The risk differences are calculated as risk in the dabigatran groups minus risk in the placebo group
Statistical Analysis 3: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.0001, normal approximation method — Multiplicity was not adjusted because of hierarchical testing from highest to lowest dose; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -32.5, 95% CI [-45.4 to -19.6] — The risk differences are calculated as risk in the dabigatran groups minus risk in the placebo group

2. Secondary Outcome: Percentage of Participants Who Have a Composite of Major VTE (Defined as Proximal DVT and PE) and VTE Related Mortality
Description: Number of participants with the composite of major VTE (defined as proximal DVT and PE) and VTE related mortality
Time Frame: 2 weeks
Population: FAS-major - FAS-major includes all patients who were randomised, treated, operated, and had an evaluable venogram for proximal DVT or confirmed symptomatic proximal DVT, PE, or VTE-related death.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 104 | 115 | 113 | 102
percentage of participants | 5.8 | 1.7 | 1.8 | 0
Statistical Analysis 1: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; Superiority of dabigatran etexilate to placebo was tested. Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Test type: Superiority or Other; p = 0.1124, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -4.0, 95% CI [-9.1 to 1.0]
Statistical Analysis 2: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.1183, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -4.0, 95% CI [-9.1 to 1.1]
Statistical Analysis 3: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p = 0.0138, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -5.8, 95% CI [-10.3 to -1.3]

3. Secondary Outcome: Percentage of Participants Who Have Proximal DVT (Deep Vein Thrombosis) During Treatment Period
Description: Number of participants who have Proximal DVT during treatment period
Time Frame: 2 weeks
Population: FAS-pDVT - FAS-pDVT includes all patients who were randomised, treated, operated, and had an evaluable venogram for proximal DVT or confirmed symptomatic proximal DVT.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 104 | 115 | 113 | 102
percentage of participants | 5.8 | 1.7 | 1.8 | 0
Statistical Analysis 1: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; Superiority of dabigatran etexilate to placebo was tested. Statistical inference was made on the basis of the normal approximation of two independent binomial distributions. The dabigatran groups were compared to the placebo group.. The null hypotheses are "Ho: placebo = 220mg", "Ho: placebo = 150mg" and "Ho: placebo = 110mg". ,All comparisons were two-sided with a significance level of 5%. Confidence intervals were two-sided with a level of 95%; Test type: Superiority or Other; p = 0.1124, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -4.0, 95% CI [-9.1 to 1.0]
Statistical Analysis 2: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.1183, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -4.0, 95% CI [-9.1 to 1.1]
Statistical Analysis 3: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0138, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -5.8, 95% CI [-10.3 to -1.3]

4. Secondary Outcome: Percentage of Participants With Symptomatic DVT (Deep Vein Thrombosis)
Description: Number of Participants expressing DVT with symptoms
Time Frame: 2 weeks
Population: FAS-op - FAS-op includes all patients who were randomly assigned to the treatment, received at least one oral dose and went through surgery.
Measure: Number; unit: Percentage of participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 124 | 133 | 126 | 129
Percentage of participants | 1.6 | 0.8 | 1.6 | 0.8
Statistical Analysis 1: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; Superiority of dabigatran etexilate to placebo was tested based on Fisher's exact test. The dabigatran groups were compared to the placebo group.. The null hypotheses are "Ho: placebo = 220mg", "Ho: placebo = 150mg" and "Ho: placebo = 110mg". ,All comparisons were two-sided with a significance level of 5%. Confidence intervals were two-sided with a level of 95%; Test type: Superiority or Other; p = 0.6107, Fisher Exact — Multiplicity was not adjusted
Statistical Analysis 2: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 1.0000, Fisher Exact — Multiplicity was not adjusted
Statistical Analysis 3: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; [analysis description as in outcome 4, analysis 1]; Test type: Superiority or Other; p = 0.6162, Fisher Exact — Multiplicity was not adjusted

5. Secondary Outcome: Percentage of Participants Who Have Total DVT (Deep Vein Thrombosis) During Treatment Period
Description: Number of participants who have Total DVT during treatment period
Time Frame: 2 weeks
Population: FAS-tDVT - FAS-tDVT includes all patients who were randomised, treated, operated, and had evaluable venogram or confirmed symptomatic DVT.
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 101 | 106 | 104 | 96
percentage of participants | 56.4 | 39.6 | 32.7 | 24.0
Statistical Analysis 1: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0155, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -16.8, 95% CI 2-sided [-30.2 to -3.4]
Statistical Analysis 2: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p = 0.0006, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -23.7, 95% CI 2-sided [-37.0 to -10.5]
Statistical Analysis 3: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority or Other; p < .0001, normal approximation method — Multiplicity was not adjusted; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Risk Difference (RD) = -32.5, 95% CI 2-sided [-45.4 to -19.6]

6. Secondary Outcome: Number of Participants With Pulmonary Embolism During Treatment Period
Description: Pulmonary embolism confirmed by pulmonary scintigraphy, pulmonary angiography or contrast CT.
Time Frame: 2 weeks
Population: FAS-op
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 124 | 133 | 126 | 129
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

7. Secondary Outcome: Number of Participants Who Died During Treatment Period
Description: All cause death, as adjudicated by the VTE events committee.
Time Frame: 2 weeks
Population: FAS-op
Measure: Number; unit: percentage of participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 124 | 133 | 126 | 129
percentage of participants | 0.0 | 0.0 | 0.0 | 0.0

8. Secondary Outcome: Number of Participants With Bleeding Events During Treatment Period
Description: Major bleeding events were defined as
  * fatal
  * clinically overt associated with loss of haemoglobin >=2g/dL in excess of what was expected
  * clinically overt leading to the transfusion of >=2 units packed cells or whole blood in excess of what was expected
  * symptomatic retroperitoneal, intracranial, intraocular or intraspinal
  * requiring treatment cessation
  * leading to re-operation
  Clinically-relevant was defined as
  * spontaneous skin hematoma >=25 cm²
  * wound hematoma >=100 cm²
  * spontaneous nose bleed >5 min
  * macroscopic hematuria spontaneous or >24 hours if associated with an intervention
  * spontaneous rectal bleeding (more than a spot on toilet paper)
  * gingival bleeding >5 min
  * any other bleeding event considered clinically relevant by the investigator
  Any bleeding events were defined as major, clinically-relevant and minor bleeding events. Minor bleeding events were defined as all other bleeding events that did not fulfil the criteria from above.
Time Frame: 2 weeks
Population: Safety set - Safety set includes all patients who were randomly assigned to the treatment, received at least one oral dose and went through surgery.
Measure: Number; unit: participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 124 | 133 | 126 | 129
participants
  Major bleeding events | 1 | 1 | 0 | 3
  Major and clinically relevant bleeding events | 4 | 1 | 1 | 5
  Any bleeding events | 10 | 13 | 13 | 14
Statistical Analysis 1: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; Comparison versus Placebo for the category major bleeding events; Test type: Superiority or Other; p = 1.0000, Fisher Exact
Statistical Analysis 2: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; Comparison versus Placebo for the category major bleeding events; Test type: Superiority or Other; p = 0.4960, Fisher Exact
Statistical Analysis 3: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; Comparison versus Placebo for the category major bleeding events; Test type: Superiority or Other; p = 0.6223, Fisher Exact
Statistical Analysis 4: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; Absolute difference versus Placebo for the category major and clinically relevant bleeding events; Test type: Superiority or Other; p = 0.1513, normal approximation method; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Absolute Difference (Percentage) = -2.5, 95% CI 2-sided [-5.9 to 1.0]
Statistical Analysis 5: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; Absolute difference versus Placebo for the category major and clinically relevant bleeding events; Test type: Superiority or Other; p = 0.1696, normal approximation method; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Absolute Difference (Percentage) = -2.4, 95% CI 2-sided [-5.9 to 1.0]
Statistical Analysis 6: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; Absolute difference versus Placebo for the category major and clinically relevant bleeding events; Test type: Superiority or Other; p = 0.7802, normal approximation method; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Absolute Difference (Percentage) = 0.7, 95% CI 2-sided [-3.9 to 5.2]
Statistical Analysis 7: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 110 mg; Absolute difference versus Placebo for the category any bleeding events; Test type: Superiority or Other; p = 0.6313, normal approximation method; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Absolute Difference (Percentage) = 1.7, 95% CI 2-sided [-5.3 to 8.7]
Statistical Analysis 8: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 150 mg; Absolute difference versus Placebo for the category any bleeding events; Test type: Superiority or Other; p = 0.5377, normal approximation method; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Absolute Difference (Percentage) = 2.3, 95% CI 2-sided [-4.9 to 9.4]
Statistical Analysis 9: Comparison: Treatment Group With Placebo vs Dabigatran Etexilate 220 mg; Absolute difference versus Placebo for the category any bleeding events; Test type: Superiority or Other; p = 0.4493, normal approximation method; Statistical inference was made on the basis of the normal approximation of two independent binomial distributions; Absolute Difference (Percentage) = 2.8, 95% CI 2-sided [-4.4 to 10.0]

9. Secondary Outcome: Blood Transfusion
Description: Blood transfusion for treated and operated patients on Day of surgery.
Time Frame: Day 0
Population: Safety set
Measure: Number; unit: participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 124 | 133 | 126 | 129
participants
  Autologous | 75 | 82 | 77 | 76
  Homologous | 5 | 4 | 4 | 2
  Autologous and homologous | 0 | 0 | 0 | 3

10. Secondary Outcome: Volume of Blood Loss
Description: Volume of blood loss for treated and operated patients during surgery.
Time Frame: Day 0
Population: Safety set
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 124 | 133 | 126 | 129
mL | 82.8 (132.0) | 90.5 (128.0) | 67.5 (96.0) | 77.3 (130.6)

11. Secondary Outcome: Laboratory Analyses
Description: Frequency of patients with possible clinically significant abnormalities.
Time Frame: First administration to end of study
Measure: Number; unit: participants
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Number analyzed (Participants) | 120 | 131 | 122 | 127
participants
  AST increase N=(120;131;122;126) | 2 | 1 | 0 | 0
  AST decrease N=(120;131;122;126) | 0 | 0 | 0 | 0
  ALT increase N=(120;131;122;126) | 2 | 0 | 1 | 0
  ALT decrease N=(120;131;122;126) | 0 | 0 | 0 | 0
  Bilirubin increase N=(120;130;122;127) | 0 | 1 | 0 | 0
  Bilirubin decrease N=(120;130;122;127) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: First administration to end of study
Arm/Group | Treatment Group With Placebo | Dabigatran Etexilate 110 mg | Dabigatran Etexilate 150 mg | Dabigatran Etexilate 220 mg
Serious Adverse Events (participants affected / at risk) | 2/124 | 3/133 | 3/126 | 2/129
Other Adverse Events (participants affected / at risk) | 62/124 | 47/133 | 60/126 | 55/129
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group With Placebo (N=124) | Dabigatran Etexilate 110 mg (N=133) | Dabigatran Etexilate 150 mg (N=126) | Dabigatran Etexilate 220 mg (N=129)
Post procedural infestation (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection bacterial (Infections and infestations) | 0 | 0 | 1 | 0
Diplegia (Nervous system disorders) | 0 | 0 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Wound haemorrhage (Vascular disorders) | 0 | 0 | 0 | 1
Haematemesis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Muscle contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Liver function test abnormal (Investigations) | 1 | 0 | 1 | 0
Wound secretion (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group With Placebo (N=124) | Dabigatran Etexilate 110 mg (N=133) | Dabigatran Etexilate 150 mg (N=126) | Dabigatran Etexilate 220 mg (N=129)
Nasopharyngitis (Infections and infestations) | 2 | 6 | 8 | 4
Insomnia (Psychiatric disorders) | 14 | 7 | 15 | 12
Headache (Nervous system disorders) | 7 | 1 | 1 | 5
Deep vein thrombosis (Vascular disorders) | 29 | 23 | 10 | 14
Constipation (Gastrointestinal disorders) | 7 | 8 | 7 | 13
Diarrhoea (Gastrointestinal disorders) | 12 | 3 | 4 | 4
Stomach discomfort (Gastrointestinal disorders) | 5 | 4 | 8 | 3
Blister (Skin and subcutaneous tissue disorders) | 7 | 5 | 10 | 8
Oedema peripheral (General disorders) | 3 | 1 | 9 | 4
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.